CLINICAL TRIAL: NCT05986851
Title: A Phase II Study to Assess Safety and Preliminary Evidence of a Therapeutic Effect of Azeliragon in Patients With MGMT Unmethylated Glioblastoma
Brief Title: Azeliragon in MGMT Unmethylated Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cantex Pharmaceuticals (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN-401
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma
Keywords: Unmethylated
MeSH Terms: conditions — Glioblastoma | interventions — azeliragon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daily oral azeliragon (Experimental): Azeliragon to be administered once daily for several days before, during, and after radiation therapy.
  Interventions: Drug: Azeliragon

INTERVENTIONS:
Drug: Azeliragon — Oral capsule

SUMMARY:
This is a phase 2 study to evaluate the safety and preliminary evidence of effectiveness of azeliragon, in combination with radiation therapy, as an initial treatment of a form of glioblastoma. Glioblastoma is a type of brain cancer that grows quickly and can invade and destroy healthy tissue. There's no cure for glioblastoma, which is also known as glioblastoma multiforme. Treatments, including surgery, radiation, and chemotherapy might slow cancer growth and reduce symptoms. New treatments of glioblastoma are needed.

DETAILED DESCRIPTION:
The study to be conducted is a phase 2 study in newly diagnosed "unmethylated" glioblastoma.

As compared to "methylated" glioblastoma "unmethylated" glioblastoma carries a worse prognosis, as it is resistant to temozolomide, the most commonly prescribed chemotherapeutic treatment. Based upon pre-clinical evidence suggesting that azeliragon may enhance the effectiveness of radiation, as well as have a delaying effect on disease progression, this study will combine daily oral azeliragon with radiation treatment, followed by continued administration of azeliragon after completion of radiation therapy.

Azeliragon is administered once daily as an oral capsule. In previous studies in patients with Alzheimer's disease and in normal volunteers, azeliragon was well tolerated for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histopathologically proven diagnosis of IDH-wildtype glioblastoma (GBM, WHO grade 4) according to the 2021 WHO classification (including subtypes such as gliosarcoma).

  2. Diagnosis must be established by open biopsy or tumor resection. Patients who have only had a stereotactic biopsy are not eligible.

  3. Supratentorial location. 4. MGMT promoter methylation is negative based on local CLIA-certified commercial laboratory tests.

  5. Must have recovered from the effects of surgery, postoperative infection, and other complications at the time the patient signs the informed consent and is determined to be eligible to participate in the study, as deemed eligible to participate per PI and sub-investigator.

  6. ≥ 18 years old. 7. Karnofsky performance status ≥ 60. 8. A diagnostic contrast-enhanced MRI or CT scan (if MRI is not available) of the brain must be performed preoperatively and postoperatively. The postoperative scan must be done within 21 days of the signing of informed consent prior to the initiation of radiotherapy. Preoperative and postoperative scans must be the same type. If CT scans were performed perioperatively, a CT should be performed before the signing of the informed consent.

  9. Study therapy must begin ≤ 7 weeks after the most recent brain tumor surgery.

  10. Adequate organ and bone marrow function as defined below:
  * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3;
  * Untransfused platelet count ≥ 75,000 cells/mm3;
  * Hemoglobin > 9.0 g/dL (Note: the use of transfusion or other intervention to achieve Hgb >9.0 g/dL is acceptable);
  * Total bilirubin ≤ 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 3x ULN 11. • Creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 mL/min using the CKD- EPI Creatinine Equation
  * If there is history of human immunodeficiency virus (HIV) infection, patients must be on effective antiretroviral therapy, and HIV viral load must be undetectable within 6 months of study enrollment.
  * If there is history of chronic hepatitis B virus (HBV) infection, patients must have either been treated or are on suppressive therapy (as indicated), and HBV viral load must be undetectable.
  * If there is history of hepatitis C virus (HCV) infection, patients must have been treated, and HCV viral load must be undetectable.

    12. Females of childbearing potential (defined as a female who is non-menopausal or surgically sterilized) must be willing to use an acceptable method of birth control (i.e., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately 13. Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form (ICF) prior to participation in any study-related activities (legally authorized representative permitted).

Exclusion Criteria:

1. Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free or not requiring active therapy for ≥ 3 years. (For example, carcinoma in situ of the breast, oral cavity, and cervix are all permissible).
2. Prior cranial RT or RT to the head and neck where potential field overlap may exist.
3. Prior use of carmustine (Gliadel) wafers or any other intratumoral or intracavitary treatment.
4. Recurrent or multicentric disease. Multicentric disease is defined as multiple discrete areas of tumor without connecting T2 signal abnormality.
5. Infratentorial disease or metastatic disease beyond the brain.
6. Known IDH mutation. IDH status could be determined by either immunohistochemistry or sequencing as evaluated per routine clinical care.
7. Patients with a serious active infection (such as a wound infection requiring parenteral antibiotics) at the time of study entry or other serious underlying medical conditions that would impair the ability of the patient to receive protocol treatment
8. Patients with any condition (e.g., psychological, geographical, etc.) that does not permit compliance with the protocol.
9. Patients receiving CYP 2C8 inhibitors noted in Section 6.3
10. Patient is unwilling or unable to comply with study procedures, including, but not limited to self-administration of oral medication
11. Patients with a gastrointestinal condition that could interfere with swallowing or absorption
12. Pregnant or breast feeding. Women of childbearing potential must a negative pregnancy test within 14 days of study entry. Females of childbearing potential who are sexually active or males with female partners of childbearing potential, where either the female or the male is unwilling to use a highly effective method of contraception during the trial and for 6 months after the last administration of azeliragon
13. Patients with concurrent participation in another interventional clinical trial or use of another investigational agent within 30 days prior to study entry. Patients who are participating in non-interventional clinical trials (e.g., QOL, imaging, observational, follow-up studies, etc.) are eligible, regardless of the timing of participation

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 2 years
  Progression-free survival (PFS) of newly diagnosed unmethylated GBM treated with the combination of RT and azeliragon.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  Overall survival (OS) of newly diagnosed unmethylated GBM after RT and azeliragon
Response rate | Up to 2 years
  To evaluate overall response rate and duration of response as per RANO criteria
Steroid requirement | Up to 2 years
  Change in requirement of dexamethasone after RT

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G Marcus, MD, Study Chair — Cantex Pharmaceuticals
Locations (8):
- United States (8):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Miami Cancer Institute - Baptist Health, Miami, Florida
  - Corewell Health, Royal Oak, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Lenox Hill Hospital, New York, New York
  - The University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - University of Utah Health Huntsman Cancer Center, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No